CLINICAL TRIAL: NCT06655493
Title: A Cross-sectional Study to Investigate Prevalence of Systemic Inflammation (hsCRP) in Cohort of Patients With HF and a Cohort of Patients With ASCVD and CKD in the Middle East
Brief Title: Levels of Inflammation in Middle East People With Cardiovascular Disease With/Without Kidney Disease
Acronym: INFLAMEAST
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8043; U1111-1303-1767 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Systemic Inflammation (hsCRP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCVD with CKD: Study participants diagnosed with Atherosclerotic Cardiovascular Disease (ASCVD) with Chronic Kidney Disease (CKD)
  Interventions: Other: No treatment given
- HFpEF or HFmrEF: Study participants diagnosed with Heart Failure (HF) with preserved ejection fraction (HFpEF) or HF with mildly reduced ejection fraction (HFmrEF)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Participants will continue their normal care and will not get any treatment as part of this study.

SUMMARY:
This study will collect medical and background information from participants with diseases that affect the heart and blood vessels (cardiovascular disease) with/without kidney disease.

The aim of the study is to assess the number of people with high levels of systemic inflammation among Middle East people with cardiovascular with/without kidney disease. Systemic inflammation means that it occurs throughout the body.

Participation in this study only requires a single visit at the clinic/hospital/medical institution. Participants will continue their normal care and will not get any treatment as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Diagnosed with ASCVD+CKD and/or HF (pEF or mrEF)

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Current participation (i.e., signed informed consent) in any other interventional clinical study.
3. Any hospitalization or unplanned visit within the last 60 days (including exacerbation of chronic disease with hospitalization).
4. Clinical evidence, or suspicion of, active infection within the last 60 days.
5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients with HF and a cohort of patients with ASCVD and CKD in the Middle East
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
High Sensitivity C-Reactive Protein (hsCRP) ≥2 mg/L | At Visit (day 0)
  Count of patients

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (20):
- Saudi Arabia (10):
  - Almoosa Specialist Hospital, Al Ahsa
  - King Fahad Armed Forces, Jeddah, Jeddah
  - King Faisal Specialist Hospital & Research Centre, Jeddah, Jeddah
  - Dr. Sulaiman Al Habib Medical Group- Olaya, Riyadh
  - King Khaled University Hospital,King Saud Univ. Med. City, Riyadh
  - Dallah Hospital_Riyadh, Riyadh
  - King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh
  - SMC, Riyadh, Riyadh
  - King Fahad Medical City, Riyadh
  - King Salman North Western Armed Force Hospital (NWAFH), Tabuk
- United Arab Emirates (10):
  - Cleveland Clinic Abu Dhabi, Abu Dhabhi
  - Tawam Hospital (SEHA), Abu Dhabhi
  - Mediclinic Abu Dhabi, Abu Dhabhi
  - Imperial college, Abu Dhabi, Abu Dhabhi
  - Tadwai hospital, Dubai
  - Rashid Hospital, Dubai
  - Dubai Hospital, Dubai
  - Fujairah Hospital, Fujairah
  - Sheikh Khalifa Hospital Fujairah, Fujairah
  - Al Qassimi Hospital, Sharjah, Sharjah city

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com